CLINICAL TRIAL: NCT00955383
Title: A Single Centre, Randomised, Double-blind, Placebo-controlled, Four-way Cross Over Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Doses of GSK2190915 in Healthy Japanese Subjects.
Brief Title: GSK2190915 Safety and Pharmacokinetic Study in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 112359
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: Japanese
MeSH Terms: conditions — Asthma | interventions — 3-(3-tert-butylsulfanyl-1-(4-(6-ethoxypyridin-3-yl)benzyl)-5-(5-methylpyridin-2-ylmethoxy)-1H-indol-2-yl)-2,2-dimethylpropionic acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- GSK2190915 (Active Comparator): GSK2190915 is a high affinity 5-lipoxygenase-activating protein (FLAP) inhibitor
  Interventions: Drug: GSK2190915
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2190915 — GSK2190915 is a high affinity 5-lipoxygenase-activating protein (FLAP) inhibitor.
  Arms: GSK2190915
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
GSK2190915 is currently in development for the treatment of asthma. This study aims to assess the safety and tolerability of single doses of GSK2190915 in healthy Japanese subjects. The study will also look at the pharmacokinetics (PK) and pharmacodynamics (PD) of single doses of GSK2190915 and aims to characterise the PK/PD relationship in healthy Japanese subjects. Twelve healthy Japanese subjects will take part in this single escalating dose study and subjects will receive one of five possible treatments, 10 mg, 50 mg, 150 mg, 450 mg GSK2190915 or placebo in each treatment period. Blood samples (for safety, pharmacokinetics and pharmacodynamics), urine samples (for safety and pharmacodynamics) and ECGs, blood pressure readings, physical examinations and a review of adverse events will take place at a number of timepoints pre and post each dose. A minimum 7 day washout between treatment periods will be required. Regardless if a subject completes or prematurely withdraws from the study, a follow up visit will be completed 7-10 days following last dose.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and 12 lead ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Japanese ethnic origin (defined as having been born in Japan with four ethnic Japanese grandparents and able to speak Japanese).
* Male or female (of non-childbearing potential) between 20 and 65 years of age inclusive, at the time of signing the informed consent. A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 of the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.

* Male subjects must agree to use one of the contraception methods listed in Section 8.1 of the protocol. This criterion must be followed from the time of the first dose of study medication until 3 months after administration of the last dose (this far exceeds the 5 half lives after administration of the last dose).
* Body weight more than or equal to 45 kg and BMI within the range 18 - 28 kg/m2 (inclusive)
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* 12 lead ECG without any clinically significant abnormality as judged by the Investigator, and QTcB or QTcF < 450 msec.
* Non-smokers (never smoked or not smoking for >6 months with <10 pack years history (Pack years = (cigarettes per day smoked/20) x number of years smoked))

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Significant cardiac, pulmonary, metabolic, renal, gastrointestinal abnormalities or other conditions that in the opinion of the investigator and/or GSK medical monitor, places the subject at an unacceptable risk as a participant in this trial.
* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines. The detection of drugs with a legitimate medical use would not necessarily be an exclusion to study participation. The detection of alcohol would not be an exclusion at screening but would need to be negative pre-dose and during the study.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including CYP3A4 inhibitors and inducers, vitamins, herbal and dietary supplements (including St John's Wort) from 14 days before screening until the follow-up visit, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. Hormone Replacement Therapy (HRT) is permitted for post-menopausal females.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500mL within a 56 day period.
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08-14 (Actual); Primary Completion 2009-10-12 (Actual); Study Completion 2009-10-12 (Actual)

PRIMARY OUTCOMES:
Clinical monitoring of blood pressure, pulse rate, ECG, physical examinations and laboratory safety data, as well as reporting of AEs. | One month following first dose.

SECONDARY OUTCOMES:
Plasma pharmacokinetic parameters including Cmax, AUC, t1/2, CL/F. | Upto 72 hours after each dose.
Leukotriene biomarkers LTB4 and LTE4 in blood and urine samples, respectively. | Upto 24 hours after each dose.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 112359 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/112359?search=study&search_terms=112359#rs
- Available data/document: Individual Participant Data Set: 112359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register